CLINICAL TRIAL: NCT06225440
Title: The Effect of Levagen+® Palmitoylethanolamide (PEA) Supplementation on Parameters of Stress, Wellbeing and Cognition in University Students
Brief Title: Impact of Levagen+® Palmitoylethanolamide (PEA) in a Cross-Over Trial Examining Stress and Cognition in University Students
Acronym: IMPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Westminster (Other)
Collaborators: Gencor Pacific Group (Industry)
Responsible Party: Principal Investigator, Mohammed Gulrez Zariwala, Professor in Translational Physiology, University of Westminster
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ETH2122-1031
Record Dates: First submitted 2024-01-03; First posted 2024-01-26 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Wellness, Psychological; Well-Being, Psychological
Keywords: nutraceutical; palmitoylethanolamide; PEA; cognition; stress; inflammation; wellness; well-being; BDNF; supplement
MeSH Terms: conditions — Psychological Well-Being; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants (and supplements) will be coded and randomly allocated (applied randomly by software) to treatment arms to eliminate order effects and maintain research staff blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levagen+® Palmitoylethanolamide (PEA) (Active Comparator): Levagen+® Palmitoylethanolamide (PEA) - 700mg/day, containing not less than 600 mg PEA.
  Interventions: Dietary Supplement: Levagen+® Palmitoylethanolamide (PEA)
- Placebo (Placebo Comparator): Placebo - Microcrystalline Cellulose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Levagen+® Palmitoylethanolamide (PEA) — Participants were instructed to swallow 2 opaque capsules (Levagen+® - 90% of PEA) with water daily at the same time of the day for 6 weeks.
  Arms: Levagen+® Palmitoylethanolamide (PEA)
Dietary Supplement: Placebo — Participants were instructed to swallow 2 opaque capsules (Microcrystalline Cellulose) with water daily at the same time of the day for 6 weeks.
  Arms: Placebo

SUMMARY:
The goal of this randomised cross-over trial is to learn about the effects of Levagen+® Palmitoylethanolamide (PEA) supplementation on cognition, wellness and well-being in young and healthy university students.

The main question it aims to answer is:

• Does the PEA supplementation affect parameters of stress, mood, cognition and well-being in university students?

Participants will complete 2 baseline on-site visits during which they will be assigned to Levagen+® Palmitoylethanolamide (PEA) treatment or placebo arm each time and:

* complete anthropometric measurements, questionnaires and surveys,
* undergo blood and saliva sampling
* complete a cognitive assessment (CANTAB)
* a randomly chosen cohort will also measure heart rate variability (HRV) over 3 days.

Researchers will compare the PEA treatment group to the placebo to see if there is a significant difference.

DETAILED DESCRIPTION:
The study will investigate the effect of Levagen+® Palmitoylethanolamide (PEA) supplementation on parameters of stress, well-being and cognition at defined time points. Assessments will be made using a combination of a range of stress measures, which will include physiological and psychometric parameters.

Physiological measures will include assessments of known biomarkers of the principal stress-sensitive physiological systems, the hypothalamic-pituitary-adrenal axis, and the autonomic nervous system, while psychometric measures will include established instruments to assess general health, somatic stress symptoms, academic stress, response to stress, cognition, and mood.

ELIGIBILITY:
Inclusion Criteria:

* Males & Females
* 18 to 40 years of age
* Fully enrolled full-time university students from London

Exclusion Criteria:

* Consumption of >14 servings of alcohol/week
* Any learning disability (e.g. dysphasia)
* Any neurobiological disorders (e.g. autism)
* Smokers Any allergies/health issues related to items being ingested
* Any serious illnesses or those on chronic medication
* Any pregnant or lactating women
* Any woman who is trying to conceive
* Any chronic gastrointestinal disorders
* Any chronic menstrual disorders (e.g. PCOS)
* Any subjects who have undergone menopause or undergoing the perimenopause transition
* Any eating disorders
* Any depression/mental disorders
* Any obese sedentary (not physically active) individual, according to BMI values
* Any abnormal blood pressure levels
* Shift work

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
To assess the influence of PEA supplementation on the perceived difficulties of test execution. | The parameters were measured during the baseline visit (day 1) and during the endpoint visit (day 42) of the 6-week supplementation period.
  Motor Screening Task (MOT) was used as a screening tool to indicate difficulties in test execution as part of the Core Cognition battery - CANTAB by Cambridge Cognition.
To assess the influence of PEA supplementation on the reaction and movement speed and attention. | The parameters were measured during the baseline visit (day 1) and during the endpoint visit (day 42) of the 6-week supplementation period.
  Reaction Time (RTI) was used to measure reaction and movement speed and attention as part of the Core Cognition battery - CANTAB by Cambridge Cognition.
To assess the influence of PEA supplementation on visual and episodic memory and visuospatial associative learning. | The parameters were measured during the baseline visit (day 1) and during the endpoint visit (day 42) of the 6-week supplementation period.
  Paired Associated Learning (PAL) was used to measure visual and episodic memory and visuospatial associative learning as part of the Core Cognition battery - CANTAB by Cambridge Cognition.
To assess the influence of PEA supplementation on short-term and spatial working memory and problem solving. | The parameters were measured during the baseline visit (day 1) and during the endpoint visit (day 42) of the 6-week supplementation period.
  Spatial Working Memory (SWM) was used to measure short-term and spatial working memory and problem solving as part of the Core Cognition battery - CANTAB by Cambridge Cognition.
To assess the influence of PEA supplementation on visual processing, recognition, and sustained attention. | The parameters were measured during the baseline visit (day 1) and during the endpoint visit (day 42) of the 6-week supplementation period.
  Rapid Visual Information Processing (RVP) was used to assess visual processing, recognition, and sustained attention as part of the Core Cognition battery - CANTAB by Cambridge Cognition.
To assess the influence of PEA supplementation on Serum Brain-derived neurotrophic factor (BDNF) levels. | The parameters were measured at the baseline visit (day 1) and at the endpoint visit (day 42) of the 6-week supplementation period.
  Serum BDNF levels were measured.

SECONDARY OUTCOMES:
To assess the influence of PEA supplementation on HRV in female population. | The parameters were measured for 3 continuous days following the baseline visit (day 1, day 2 and day 3) and for 3 continuous days following the endpoint visit (day 42, day 43 and day 44) of the study period.
  HRV was measured for 3 full days.
To study the influence of PEA supplementation on the degree of perceived stress in females. | The parameters were measured for 3 continuous days following the baseline visit (day 1, day 2 and day 3) and for 3 continuous days following the endpoint visit (day 42, day 43 and day 44) of the study period.
  The Perceived Stress Scale (PSS) a 10-item questionnaire was used to measure the degree to which situations in the participant's life were appraised as stressful.
  The questions investigate how often certain feelings and thoughts were experienced on a five-point scale from 'never' to 'very often' (never =0, almost never = 1, sometimes = 2, fairly often = 3 and very often = 4) during the 3-day observation periods. To calculate a total PSS score, responses to the four positively stated items (items 4, 5, 7 and 8) first need to be reversed (i.e. 0 => 4; 1 => 3; 2 => 2; 3 => 1; 4 => 0).
  The PSS score were then obtained by summing across all items. Higher scores indicate higher levels of perceived stress.
To study the influence of PEA supplementation on perceived emotions in females. | The parameters were measured for 3 continuous days following the baseline visit (day 1, day 2 and day 3) and for 3 continuous days following the endpoint visit (day 42, day 43 and day 44) of the study period.
  The Positive and Negative Affect Schedule (PANAS) was used to assess feelings of both positive and negative emotions experienced simultaneously.
To study the influence of PEA supplementation on well-being in females. | The parameters were measured for 3 continuous days following the baseline visit (day 1, day 2 and day 3) and for 3 continuous days following the endpoint visit (day 42, day 43 and day 44) of the study period.
  Student Well-being Process Questionnaire (WPQ) a 44-item questionnaire was used to examine predictors of positive well-being, adverse mental health, and cognitive function. The responses to questions 1 - 42 were assessed on a 10-point scale and or questions 43 and 44 on a 4-point scale. Where with outcomes related to positive well-being high scores = more positive; with outcomes related to adverse mental health high scores = more negative and with outcomes related to cognitive function high scores = more cognitive problems. Positive well-being was predicted by high positive personality, high social support and low stressor and low negative coping scores. Negative outcomes were predicted by high stressor, coping and conscientiousness scores, and low positive personality and low social support scores. Cognitive problems were predicted by high stressor and negative coping scores and low positive personality scores.
To assess the influence of PEA supplementation on parameters of inflammation. | The parameters were measured at the baseline visit (day 1) and at the endpoint visit (day 42) of the 6-week supplementation period.
  Interferon-gamma (pg/mL), Interleukin-1 beta (pg/mL), Interleukin 6 (pg/mL), Interleukin 10 (pg/mL), Tumour necrosis factor alpha (pg/mL) levels were measured.
To assess the influence of PEA supplementation on Salivary Cortisol | The parameters were measured in morning and afternoon samples collected over 3 continuous days following the baseline visit (day 1, day 2 and day 3) and 3 continuous days following the endpoint visit (day 42, day 43 and day 44) of the study period.
  Salivary Cortisol levels were measured during morning, afternoon and evening for 3 days following each baseline and endpoint visit at home.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Gulrez Zariwala, PhD, Principal Investigator — University of Westminster; Sanjoy Deb, PhD, Principal Investigator — Anglia Ruskin University
Locations (1):
- University of Westminster, London, United Kingdom

REFERENCES:
- [Derived] Deb SK, Kim N, Parolin B, Renshaw D, Zariwala MG. The effects of formulated palmitoylethanolamide supplementation on indicators of stress and heart rate variability in female university students: a randomised cross-over trial. Front Nutr. 2025 Sep 19;12:1586409. doi: 10.3389/fnut.2025.1586409. eCollection 2025. PMID 41049366